CLINICAL TRIAL: NCT00004142
Title: Phase II Study of Radiofrequency Ablation of Colorectal Cancer Liver Metastases Combined With Post-Ablation Hepatic Arterial Infusion of Floxuridine Alternating With 5-Fluorouracil
Brief Title: Radiofrequency Ablation Followed By Hepatic Artery Chemotherapy in Treating Patients With Colorectal Cancer That Has Spread to the Liver
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ID98-035; P30CA016672 (NIH); MDA-ID-98035 (Other: UT MD Anderson Cancer Center); NCI-G99-1616; CDR0000067373 (Registry Identifier: NCI PDQ)
Record Dates: First submitted 1999-12-10; First posted 2004-03-15 (Estimated); Last update posted 2018-10-26 (Actual); Status verified 2018-10

CONDITIONS: Colorectal Cancer; Metastatic Cancer
Keywords: stage IV colon cancer; stage IV rectal cancer; recurrent colon cancer; recurrent rectal cancer; liver metastases
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasm Metastasis; Colonic Neoplasms; Rectal Neoplasms | interventions — Floxuridine; Fluorouracil; Radiofrequency Ablation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Radiofrequency Ablation + HAI of Floxuridine/5-FU (Experimental): Radiofrequency Ablation Combined With Post-Ablation Hepatic Arterial Infusion (HAI) of Floxuridine Alternating With 5-Fluorouracil (5-FU)
  Interventions: Drug: Floxuridine; Drug: Fluorouracil (5-FU); Procedure: Conventional surgery; Procedure: Radiofrequency ablation

INTERVENTIONS:
Drug: Floxuridine — Part of hepatic arterial chemotherapy on days 1-7. Treatment repeats every 5 weeks for 6 courses.
Drug: Fluorouracil (5-FU) — Part of hepatic arterial chemotherapy over 1 hour on days 15, 22, and 29. Treatment repeats every 5 weeks for 6 courses.
  Other Names: 5-FU; 5-Fluorouracil; Adrucil; Efudex
Procedure: Conventional surgery — Open laparotomy to identify target tumor in liver using intraoperative ultrasound.
  Other Names: open laparotomy
Procedure: Radiofrequency ablation — Radiofrequency tissue ablation over 20 minutes to each tumor.

SUMMARY:
RATIONALE: Radiofrequency ablation may be able to shrink or destroy cancer cells. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Chemotherapy delivered directly into the blood vessels of the liver may prevent new tumors from growing. Combining these therapies may be an effective treatment for colorectal cancer that has spread to the liver.

PURPOSE: Phase II trial to study the effectiveness of radiofrequency ablation followed by chemotherapy delivered directly into the blood vessels of the liver in treating patients who have colorectal cancer that has spread to the liver.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the safety and efficacy of radiofrequency tissue ablation followed by hepatic arterial chemotherapy with floxuridine and fluorouracil in patients with colorectal cancer metastatic to the liver.

OUTLINE: Patients undergo an open laparotomy to identify the target tumor in the liver using intraoperative ultrasound followed by radiofrequency tissue ablation over 20 minutes to each tumor and placement of hepatic arterial catheter. Within 35 days postoperatively, patients receive hepatic arterial chemotherapy consisting of floxuridine on days 1-7 and fluorouracil over 1 hour on days 15, 22, and 29. Treatment repeats every 5 weeks for 6 courses. Patients are followed at 1 month, every 3 months for 2 years, every 6 months for 3 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 42 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed colorectal cancer metastatic to the liver No preoperative or intraoperative evidence of extrahepatic metastasis including clinical, radiographic, gross or microscopic evidence Tumors must be no more than 4 cm in diameter No more than 6 total tumors May have failed prior systemic chemotherapy Failure of 1 prior intra-arterial regimen excluding floxuridine, fluorouracil, or another fluoropyrimidine allowed if liver enzymes recovered No evidence of cirrhosis No gross ascites

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: Zubrod 0-2 Life expectancy: At least 16 weeks Hematopoietic: Granulocyte count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin no greater than 1.5 mg/dL Renal: Creatinine no greater than 1.5 mg/dL OR Creatinine clearance at least 60 mL/min Other: No active duodenal or gastric ulcers Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: See Disease Characteristics At least 4 weeks since prior chemotherapy (6-8 weeks since nitrosoureas or mitomycin) Endocrine therapy: Not specified Radiotherapy: At least 4 weeks since prior radiotherapy No prior radiotherapy to the liver Surgery: Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 1998-08-05 (Actual); Primary Completion 2003-12-09 (Actual); Study Completion 2003-12-09 (Actual)

PRIMARY OUTCOMES:
Patient Tumor Response Rate | At 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Lee M. Ellis, MD, Study Chair — M.D. Anderson Cancer Center
Locations (1):
- University of Texas - MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center Website — http://www.mdanderson.org